CLINICAL TRIAL: NCT00696397
Title: Sleep Disturbance in Atopic Dermatitis: A Comprehensive Investigation of Opiates, Neuropeptides, Barrier Function, Scratching and Sleep Physiology
Brief Title: Comprehensive Investigation of Opiates, Neuropeptides, Barrier Function, Scratching and Sleep Physiology
Status: Completed | Type: Observational
Sponsor: Wake Forest University (Other)
Responsible Party: Sponsor
Organization: Wake Forest University Health Sciences (Other)
Other Study IDs: 00000046
Record Dates: First submitted 2008-06-09; First posted 2008-06-12 (Estimated); Last update posted 2017-03-16 (Actual); Status verified 2012-08

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, dermal microdialysate
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A: adult men and women between 18 and 50 years of age with atopic dermatitis

SUMMARY:
The purpose of this research is to study the sleep patterns of people with moderate to severe atopic dermatitis and how itching affects those patterns. This study will also measure your body's activity during sleep using non-invasive tests described below.

ELIGIBILITY:
Inclusion Criteria:

* Adult men and women who are between 18 and 50 years of age
* Diagnosis of moderate to severe atopic dermatitis including involvement of the forearm confirmed by published consensus diagnostic criteria57 (except for healthy control subjects)
* Subjects must be in general good health with no other skin disease, disease state or physical condition which would impair evaluation of their skin or which would increase their health risk by study participation
* Subjects must be willing to stay overnight in the sleep laboratory and/or to undergo dermal microdialysis
* Women of child bearing age will be required to have a negative pregnancy test in order to enroll in the study and will be required to maintain adequate birth control throughout the study.

Exclusion Criteria:

* Adults over age 50
* Children less than 18 years of age.
* Unable to complete the required measures
* Diagnosis with other skin diseases that would affect the measurement of transepidermal water loss (TEWL) as determined by the investigators
* Currently enrolled in any investigational study in which the subject is receiving any type of drug, biologic, or non-drug therapy and patients undergoing treatment with another investigational drug or approved therapy for investigational use within 28 days prior to study participation
* Evidence of depression based on the Beck Depression Inventory (BDI > 10)
* Evidence of sleep apnea based on the results of the Epworth Sleepiness Scale score (ESS > 10)
* Evidence of insomnia based on the Insomnia Severity Index (ISI) that is determined by the principal investigator to be unrelated to atopic dermatitis
* Individuals who work shifts between 8 pm and 6 am because such night shifts can alter subjects' circadian rhythms.
* Typically sleep less than 5 hours per night
* Reported habitual bedtime earlier than 9pm or later than 1 am (> 2 times per week on screening diaries)
* Reported habitual rising time later than 9 am (> 2 times per week on screening diaries
* Diagnosis of sleep apnea, periodic limb movement disorder, or restless leg syndrome 58
* Consumption of more than 3 alcoholic beverages per day
* Consumption of more than 4 caffeinated beverages per day 59-61
* Chronic pain judged to be a significant sleep-disturbing factor as determined by the investigators62
* Current treatment with lipophilic beta blockers, opioids, glucocorticoids, theophylline, or other medications known to interfere with sleep as determined by the investigators 63-69
* Uncontrolled asthma or COPD 70-73
* Uncontrolled thyroid disease 74,75
* Poorly controlled diabetes mellitus
* Poorly compensated congestive heart failure 76
* Use of herbal or naturopathic treatments for sleep
* Habitual smoking between 11 pm and 7 am 77,78
* Use of illicit drugs

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: adult men and women between 18 and 50 years of age with atopic dermatitis
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2006-03; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
To assess whether there are differences in dermal and serum opiate levels and neuropeptides involved in atopic dermatitis between day and night | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Gil Yosipovitch, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences Dermatology, Winston-Salem, North Carolina, United States